CLINICAL TRIAL: NCT04269135
Title: Preschool Children: Fit, Healthy and Smart: PREFIT-Chile - Study Linking Physical Fitness to Non Invasive Health-Related Markers and Executive Function
Brief Title: Fit, Healthy and Smart Preschool Children: PREFIT-Chile
Acronym: PREFIT-Chile
Status: Completed | Type: Observational
Sponsor: Playa Ancha University (Other)
Collaborators: University of Chile (Other); Universidad de Granada (Other)
Responsible Party: Principal Investigator, Johana Soto Sánchez, Physical Education Teacher, Playa Ancha University
Other Study IDs: REDI 170474
Record Dates: First submitted 2020-02-07; First posted 2020-02-13 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Child, Preschool
Keywords: Physical fitness; Risk factors; Anthropometrics; Blood pressure; Neuropsychological Tests; Physical activity; Motor skills
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Investigating the interrelationship between physical condition, non-invasive health markers and executive function in preschoolers, is based on the current health and cognitive development situation of this population, especially the low socioeconomic level. National figures estimate that the prevalence of overweight / obesity in the preschool population reaches 53.6%, exposing not only the development of cardiovascular and metabolic diseases, but also affect cognitive potential.

Physical condition is a powerful health marker independent of nutritional status. Its evaluation together with the evaluation of non-invasive health markers and executive function in preschoolers inside educational establishments is essential to investigate alterations at an early age that could be prevented with adequate interventions in schools. However, to achieve this, valid, reliable and comparable tools are needed internationally.

Objective: to analyze the factors that affect the configuration of a diagnostic model which includes the physical fitness and physical activity levels, motor development, non-invasive risk factors and neuropsychological development in preschoolers.

Methods: Observational study, case only, cross sectional. Enrollment 544 preschool child 4 to 5 years old. Primary Outcome is Physical fitness to "Prefit Battery", Secondary outcome non-invasive risk factors (Blood pressure, BMI, Waist circumference, neck circumference) Physical activity, Motor skills and Neuropsychological development.

expected results: Determine the degree of association of physical fitness with non-invasive risk factors and neuropsychological development in preschoolers, determine the influence that physical activity level and motor development have on physical fitness and development a diagnostic model which includes the physical fitness and physical activity levels, motor development, non-invasive risk factors and neuropsychological development in Chilean preschoolers.

DETAILED DESCRIPTION:
In recent years it has been demonstrated that physical fitness , which is linked to a higher level of physical activity has a positive effect on the health status of adults, adolescents and children, especially by lowering the probability of developing overweight and/or obesity. At the same time, recent research has shown that there is a positive relationship between fitness with brain structure and executive function in children.

In Chile, overweight and obesity constitute a public health problem in children. National figures show that the prevalence of overweight / obesity among preschool children reached 53.6% in 2018 exposing the children not only the development of cardiovascular and metabolic diseases , but also affecting motor and cognitive development. Obesity has been shown to influence a country´s economic development, such as salary and productivity. The Economic Commission for Latin America and the Caribbean in 2017 determined that the health cost derived from obesity In Chile was equivalent to 0,2% of the national Gross Domestic Product. It is expected that by 2078, the estimated annual cost produced by an increasing prevalence overweight / obesity will be approximately 1 billion dollars.

Because it is not economically viable in Chile to determine in every overweight/obese child the probability of developing chronic diseases later in life, it is of utmost importance to have valid, simple and reliable indicators to discriminate at an early age, children that are at greatest risk. In this respect, physical fitness appears as a powerful health marker independent of the nutritional status. Evaluation of fitness as well as that of non-invasive health markers, motor development and neuropsychological development in preschool children in schools, constitute an excellent opportunity to investigate at an early age, alterations that could be prevented with adequate interventions in schools that would probably be significantly less costly than interventions applied later on. To achieve this goal, valid and reliable tools have to be developed that are also comparable with similar ones developed elsewhere.

With this background, The research objective is to analyze the factors that affect the configuration of a diagnostic model which includes the physical fitness and physical activity levels, motor development, non-invasive risk factors and neuropsychological development in preschoolers.

The hypothesis is that there is a positive association between physical fitness, non-invasive health markers and neuropsychological functions in preschool children, thus enabling to generate a predictive diagnostic model based on physical fitness.

1. The primary outcome is to determine the degree of association of physical fitness with non-invasive risk factors and neuropsychological development in preschoolers
2. The second outcome is to determine the influence that physical activity level and motor development have on physical fitness among preschool children.

This research aims a) to establish that physical fitness in preschool children may be considered as a diagnostic tool of the health status of children (independent of their nutritional status), and b) to determine the possible impact that the physical fitness level has on neuropsychological development

ELIGIBILITY:
Inclusion Criteria:

* Preschool child, 4 to 5 years old, Speaking Spanish and Agree to the commitment

Exclusion Criteria:

* Chronic pediatric disease (except for obesity) Cardiovascular or metabolic disease, neurological, respiratory bronchial disease and Orthopedic limitation.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preschoolers from 4 to 5 years old, incorporated into the school system and attending kindergartens and schools, residents of the central area of Chile, to detail IV region of "Coquimbo", V region of "Valparaíso", VI region of the "Liberator Bernardo O'Higgins" and the "Metropolitan" Region
Sampling Method: Non-Probability Sample
Enrollment: 868 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Measurement of "Physical fitness" | "1 Day" on "45 minute"
  Results from PREFIT battery; is composed of the following tests: the 20 m shuttle-run test for assessing cardiorespiratory fitness, the handgrip-strength and the standing long-jump tests for assessing muscular musculoskeletal fitness, and the 4x10 m shuttle-run.

SECONDARY OUTCOMES:
Measurement "Blood Pressure" | "1 Day" on "15 minutes"
  Measured in the right arm, The child stay a quiet for 3-5 min before measurement, with the back supported and feet uncrossed on the floor.
Estimated "Body Mass Index" | "1 Day" on "10 minute"
  Measured the weight (kg) and Height (m), then applicate the equation weight/height^2 to determinate de value.
Measurement "Waist circumference" | "1 Day" on "10 minutes"
  The child stands erect with the abdomen relaxed, the arms at the sides and the feet together. The tester faces the child and places an inelastic tape around him / her, in a horizontal plane, The measurement will be made at the level of the navel and so that the tape forms a horizontal plane parallel to the ground.
Measurement "neck circumference" | "1 Day" on "10 minute"
  The child stands tall, arms at the sides and feet together. The tester looks at the Child and places an inelastic tape around of thyroid cartilage
Measurement "Physical activity" | "7 Days"
  The equipment will be located in the right hip area with an adjustable elastic belt. Record the information with an interval of 15 seconds (time) with a frequency of 100 Hz, the above is executed by means of the Actilife-6 software
Measurement "Motor Skills" | "1 Day" "45 minutes"
  the standardized instrument called Test of Gross Motor Development (TGMD-2) will be used. Which measures 12 gross motor skills
Measurement "Neuropsychological development" | "1Day" "30 minutes"
  It will be evaluated by means of standardized tests, battery of child computerized neuropsychological evaluation (BENCI), which requires children to perform a series of activities on an iPad, where the following functions will be evaluated: Visomotor coordination, Processing speed, Language and Executive function (only in 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Johana P Soto-Sánchez, PhD, Principal Investigator — Playa Ancha University
Locations (1):
- Playa Ancha University, Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burkhalter TM, Hillman CH. A narrative review of physical activity, nutrition, and obesity to cognition and scholastic performance across the human lifespan. Adv Nutr. 2011 Mar;2(2):201S-6S. doi: 10.3945/an.111.000331. Epub 2011 Mar 10. PMID 22332052
- [Result] Chaddock-Heyman L, Erickson KI, Holtrop JL, Voss MW, Pontifex MB, Raine LB, Hillman CH, Kramer AF. Aerobic fitness is associated with greater white matter integrity in children. Front Hum Neurosci. 2014 Aug 19;8:584. doi: 10.3389/fnhum.2014.00584. eCollection 2014. PMID 25191243
- [Result] Chaddock-Heyman L, Hillman CH, Cohen NJ, Kramer AF. III. The importance of physical activity and aerobic fitness for cognitive control and memory in children. Monogr Soc Res Child Dev. 2014 Dec;79(4):25-50. doi: 10.1111/mono.12129. PMID 25387414
- [Result] Junta Nacional Escolar de Auxilio y Becas (JUNAEB). Informe Mapa Nutricional 2018 de Chile. Lira, M. 2019
- [Result] Fernández, A., Martínez, R., Carrasco, I., & Palma, A. (2017). Impacto social y económico de la malnutrición: modelo de análisis y estudio piloto en Chile, el Ecuador y México. Retrieved from https://www.cepal.org/es/publicaciones/41247-impacto-social-economico-la-malnutricion-modelo-analisis-estudio-piloto-chile
- [Result] Ortega FB, Cadenas-Sanchez C, Sanchez-Delgado G, Mora-Gonzalez J, Martinez-Tellez B, Artero EG, Castro-Pinero J, Labayen I, Chillon P, Lof M, Ruiz JR. Systematic review and proposal of a field-based physical fitness-test battery in preschool children: the PREFIT battery. Sports Med. 2015 Apr;45(4):533-55. doi: 10.1007/s40279-014-0281-8. PMID 25370201
- [Derived] Soto-Sanchez J, Leyton-Dinamarca B, Kain J, Fernandez-Valero P, Castro-Cisterna S, Arias-Tellez MJ, Ortega FB. Reliability of the PREFIT fitness-test battery in Chilean preschoolers. Front Pediatr. 2026 Jan 12;13:1654731. doi: 10.3389/fped.2025.1654731. eCollection 2025. PMID 41602872